CLINICAL TRIAL: NCT04485676
Title: Dalbavancin in Real Clinical Practice in Spain: a Two-year Retrospective Study
Brief Title: Dalbavancin in Real Clinical Practice in Spain
Acronym: REAL-DAL
Status: Completed | Type: Observational
Sponsor: Angelini Farmacéutica (Industry)
Collaborators: Effice Servicios Para la Investigacion S.L. (Industry)
Responsible Party: Sponsor
Other Study IDs: ANG-DAL-2019-01
Record Dates: First submitted 2020-06-16; First posted 2020-07-24 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2021-05

CONDITIONS: Skin Diseases, Bacterial; Skin Diseases, Infectious
MeSH Terms: conditions — Skin Diseases, Bacterial; Skin Diseases, Infectious

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Dalbavancin: Patients to be included in this study have been treated with Dalbavancin according to clinician's judgement and clinical practice according national or international guidelines.
  Dalbavancin is indicated for the treatment of acute bacterial skin and skin structure infections (ABSSSI) in adults. Information about dosing treatment will be collected.

SUMMARY:
The aim of this study is to describe the real clinical use of Dalbavancin in Spain between January 2018 and December 2019.

DETAILED DESCRIPTION:
Dalbavancin is a new lipoglycopeptide approved for the treatment of ABSSSIs (Acute Bacterial Skin and Skin-Structure Infections) with activity against Gram-positive pathogens, including MRSA. Dalbavancin has unique pharmacokinetics properties, with a terminal half-life of 14.4 days, permitting a single intravenous dosing. Dalbavancin has shown a favourable efficacy and safety profile in patients with ABSSSI in randomized controlled trials. However, information regarding daily clinical practice is limited. The main objective of this study is to describe the real clinical practice with Dalbavancin in Spain.

ELIGIBILITY:
Inclusion Criteria:

1. Adult man and woman (≥ 18 years) at the time of receiving dalbavancin
2. Patients receiving at least one dose of dalbavancin between 1st January 2018 and 31st December 2019
3. Patients with medical follow-up information registered in clinical records for about 90 days after completing the treatment
4. Written informed consent requested according to local regulation, IEC and protocol requirements

Exclusion Criteria:

1. Patient enrolled in a clinical trial in which treatment with dalbavancin is managed through a protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with dalbavancin from 1st January 2018 to 31st December 2019
Sampling Method: Non-Probability Sample
Enrollment: 187 (Actual)
Dates: Start 2020-07-15 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-02-21 (Actual)

PRIMARY OUTCOMES:
Demographic and clinical characteristics of patients treated with dalbavancin | patients treated with dalbavancin between January 2018 and December 2019
  To describe the demographic and clinical characteristics of patients treated with dalbavancin (primary objective)
Variables related to dalbavancin treatment | patients treated with dalbavancin between January 2018 and December 2019
  To describe the demographic and clinical characteristics of patients treated with dalbavancin (primary objective)

SECONDARY OUTCOMES:
Effectiveness/Clinical response | From 48-72h after the end of treatment until 90 days after last dose of dalbavancin
  Clinical response (signs and symptoms) evaluated at the end of treatment
Effectiveness/Relapse | 90 days after after last dose of dalbavancin
  Relapse (Yes/No)
Safety. Adverse events | From first dose until 90 days after last dose of dalbavancin
  Rate of adverse events Rate of treatment discontinuation due to Adverse events
Treatment compliance | : From first dose until 90 days after last dose of dalbavancin
  Patient received the full dose of dalbavancin (Yes/No)
Doctors opinion on infection management with dalbavancin (1) | From first dose until 90 days after last dose of dalbavancin
  Degree of physician satisfaction on management with dalbavancin: Dissatisfied, Little satisfied, Satisfied, Very satisfied
Doctors opinion on infection management with dalbavancin (2) | From first dose until 90 days after last dose of dalbavancin
  Physician assessment on potential reduction in the number of days of hospital stay (Yes/No)

CONTACTS AND LOCATIONS:
Overall Officials: Benito Almirante, PhD, Principal Investigator — Hospital Vall d'Hebrón
Locations (7):
- Spain (7):
  - Hospital Universitario A Coruña, A Coruña
  - Hospital Universitari Vall d'Hebrón, Barcelona
  - Hospital Clínic Barcelona, Barcelona
  - Hospital Universitario Virgen de las Nieves, Granada
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universtario La Fe, Valencia